CLINICAL TRIAL: NCT06976801
Title: Prospective, Randomized-control Trial Comparing Standard Intramedullary Tibial Fixation With Micromotion Tibial Intramedullary Fixation
Brief Title: Tibial IMN Vs. Tibial Micromotion IMN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-0601
Record Dates: First submitted 2025-01-13; First posted 2025-05-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-05

CONDITIONS: Tibial Fracture
Keywords: Unstable tibial fracture; intramedullary nail; micromotion tibial nail fixation
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Intervention Model Description: The only intervention involved in this study is randomization between the two surgical devices. Subgroups will be determined using equal block randomization. Block randomization will be used for this study. Blocks will be set to groups of 4 with each block of 4 comprising 2 MMIMNF and 2 IMNF opaque envelopes in random order. The envelope will be opened in the OR prior to beginning the procedure. This ensures subjects are blinded to their initial treatment modality. Standard of care will be followed for all clinical decisions beyond the type of surgical procedure to be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- micromotion tibial intramedullary fixation (Experimental): Subject will receive micromotion tibial intramedullary fixation
  Interventions: Device: Intramedullary tibial Nail
- non-micromotion tibial nail fixation (Active Comparator): Subject will receive non-micromotion tibial nail fixation
  Interventions: Device: Intermedullary nail

INTERVENTIONS:
Device: Intramedullary tibial Nail — Subjects will receive the micromotion MicroMotion Intramedullary tibial Nail
  Other Names: MicroMotion Intramedullary tibial Nail
  Arms: micromotion tibial intramedullary fixation
Device: Intermedullary nail — The non-micromotion intermedullary nail
  Arms: non-micromotion tibial nail fixation

SUMMARY:
Our null hypothesis is that micromotion tibial intramedullary fixation (IMFN) does not impact union or complication rates when compared to standard of care treatment with non-micromotion tibial nail fixation. There are no current or past randomized controlled trials comparing these fixation techniques to one another. There is good data supporting both the use of intramedullary fixation for tibial fractures alone, and in high-risk patient populations (open fractures, GSW tibial fractures). However, the effectiveness of these methods with respect to each other has never been investigated. The knowledge gained will allow us to potentially influence and adapt protocols to treat this patient population. Additionally, resources available at our institution provide a supportive framework with which to maintain contact with patients after hospital discharge. These key factors will allow us to perform a robust analysis of this population, to include outcomes measures of function and complications.

With much of the limited existing literature on tibial nails being in very defined populations, without a strong comparison group there is no clear guidance on when the use of a micromotion device is indicated. Our approach to randomize our patients will reduce the bias that exists in the current literature and provide a robust spectrum of injuries to sub analyze and compare.

Objectives Primary Objective Compare post-operative union rates in tibial shaft patients treated with 2 types of intramedullary rod fixation devices.

Secondary Objective(s) Compare complication rates, patient reported outcomes, range of motion, pain and radiographic/sonographic outcomes in patients treated with tibial nails.

DETAILED DESCRIPTION:
The advent of the intramedullary nail (IMN) has revolutionized the treatment of tibial shaft fractures due to its percutaneous route of insertion, frequent facilitation of immediate weightbearing, and high rate of union. Recent research has revealed that selection of an appropriate IMN diameter is vital for maintaining fracture reduction and preventing complications. Using a larger diameter nail increases construct stability, permits load-sharing, and may lead to higher rates of union. On the other hand, aggressive reaming to permit a larger nail diameter can result in iatrogenic fracture upon insertion or removal.

Modern tibial nail designs have remained largely unchanged in the last 20 years with small ergonomic and efficiency changes without large scale improvements in their biomechanical induction of bone healing at the fracture site. Traditionally they include distal locking screws as well as proximal locking screws that are either fixed or dynamic allowing for small but largely irrelevant amounts of motion. Our understanding of bone healing and indirect bone generation includes the concept of micromotion which induces the creation of fibrous followed by bony callus. This concept requires strain levels and adequate micromotion at fracture sites to be biomechanically advantageous. One new tibial nail device recently available in the US and FDA approved for tibial nail fixation hopes to improve the biomechanical and biology environment for tibial healing, the OrthoXel tibial nail system. Unfortunately, there is a paucity of strong clinical data to support it. Additionally, there have been no prospective, randomized studies investigating the used of this nail compared to standard tibial nail designs and no studies have evaluated it in high risk tibial non-union patients..

The primary purpose of this study is to perform a high-quality randomized control trial comparing intramedullary tibial nail fixation with standard design nails compared to a micromotion tibial nail device to evaluate the rates of union and post-operative outcomes. In an evaluation of patient factors, fracture patterns and patient reported outcomes, the investigators will bring clarity to the question of indications for the micromotion tibial nail in standard and high risk patients. To characterize our patient population, the investigators will evaluate type of injury (closed, open, gunshot wound), fracture morphology (OTA classification), patient risk factors (age, isolated vs. poly-trauma, Comorbidities, smoking, and Vit D levels) and surgical outcomes (blood loss, surgical time, construct stability). In addition to objective radiographic, ultrasonographic and physical exam outcomes, the investigators will collect patient reported outcomes in the form of PROMIS CAT and VAS scores.

Given the existing limitations in the literature, there is no guidance on indications for use of micromotion tibial nail fixation (MMIMNF) compared to standard intramedullary nail fixation (IMNF). By taking an approach that will be prospective and randomized, while assessing all known risk factors, the investigators expect our results will guide surgical treatment decisions around the use of these devices and in which populations they may be most useful. .

The proposed trial will be a parallel-group, superiority trial with equal randomization enrolling 242 tibial nail patients. Patients will be categorized into 2 cohorts: IMNF fixation(cohort 1), and MicroMotion Intramedullary tibial Nail fixation (cohort 2). The primary outcome will be nonunion. Secondary outcomes will include: overall complications (as a composite result (Infection ((deep and superficial)), revision surgery rate, removal of metalwork, non-union, malunion, amputation and death). Patient-Reported Outcomes Measurement Information System Physical Function Computerized Adaptive Testing (PROMIS PT CAT) scores, range of motion (ROM), pain, radiographic outcomes, time to bridging callus based on mRUST (>11) on Xray, time to single leg stance, and degree of callus seen on ultrasound at 6 & 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Unstable tibial fracture recommended for surgical intervention

Exclusion Criteria:

1. Patients not meeting inclusion criteria (Stable fracture patterns)
2. Previously non-ambulatory patients
3. Delayed presentation of fracture (>4 weeks)
4. Fractures that the treating surgeon indicates requires additional fixation strategies to achieve stability
5. Patients with an active infection or wound at the surgical site
6. Utilizing worker's compensation at the time of screening
7. Any previous ligament or fracture surgery on the index site
8. Inflammatory rheumatic disease or other rheumatic disease
9. Immune compromised patients (hepatitis, HIV, etc.)
10. Non-English-speaking patients
11. Unwilling or unable to participate or follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Compare post-operative union rates | six months
  Compare post-operative union rates in tibial shaft patients treated with 2 types of intramedullary rod fixation devices.

SECONDARY OUTCOMES:
Compare complication rates | one year
  Compare complication rates outcomes in patients treated with tibial nails
Time to single leg stance | one year
  Time (in days) it takes for the subject stand on a single leg.
Any difference in patient reported outcomes scores physical function | one year
  Patient Reported outcome scores physical function scores are reported on a T-score scale that ranges from 20-80, with higher scores indicating greater physical function.
Any difference in patient reported outcomes scores pain interference | one year
  Patient Reported outcome scores pain interference scores are reported on a T-score scale that ranges from 6-30, with higher scores indicating greater physical function.
Ultra sound callus | 6 weeks
  Checking if a callus has appeared
Ultra sound callus | 12 weeks
  Checking if callus has appeared
Visual analog pain scale score | one year
  Visual analog pain scale scores for the subject. Scored on a scale of 0 - 10. 0 no pain and 10 worst pain.

OTHER OUTCOMES:
Smoking Status | one year
  Comparing the smoking status (yes/no and pack years) and return to OR timelines
Visual analog pain scale score | one year
  Visual analog pain scale score? 0 (no pain) - 10 (worst pain)
Fixation failure rate | one year
  Comparing the fixation failure rates between the two groups and return to OR timelines
Radiographic Mal-union | one year
  Comparing Radiographic Mal-union rates between groups
Radiographic Non-union | one year
  Comparing rates Radiographic Non-union between groups
Any difference in Patient reported outcomes scores depression | one year
  Patient Reported outcome scores depression scores are reported on a T-score scale that ranges from 8 - 40, with higher scores indicating greater depression.
Reoperation Rate | one year
  Comparing Reoperation Rate between groups
Any difference in Patient reported outcomes scores anxiety | one year
  Patient Reported outcome scores anxiety scores are reported on a T-score scale that ranges from 7 - 35, with higher scores indicating greater anxiety.
Infection Rate (Superficial and Deep) | one year
  Comparing Infection Rate (Superficial and Deep) between group
Amputation Ratee | one year
  Comparing Amputation Rate between groups
Knee & ankle Range of Motion | one year
  Comparing Knee & ankle Range of Motion between groups
Diabetes | one year
  Comparing diabetes between subjects and return to OR timelines
BMI | one year
  Comparing BMI in subjects and and return to OR timelines

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Background] Whittle AP, Wester W, Russell TA. Fatigue failure in small diameter tibial nails. Clin Orthop Relat Res. 1995 Jun;(315):119-28. PMID 7634660
- [Background] Hutson JJ, Zych GA, Cole JD, Johnson KD, Ostermann P, Milne EL, Latta L. Mechanical failures of intramedullary tibial nails applied without reaming. Clin Orthop Relat Res. 1995 Jun;(315):129-37. PMID 7634661
- [Background] Bonafede M, Espindle D, Bower AG. The direct and indirect costs of long bone fractures in a working age US population. J Med Econ. 2013;16(1):169-78. doi: 10.3111/13696998.2012.737391. Epub 2012 Oct 22. PMID 23035626
- [Background] Weber CD, Hildebrand F, Kobbe P, Lefering R, Sellei RM, Pape HC; TraumaRegister DGU. Epidemiology of open tibia fractures in a population-based database: update on current risk factors and clinical implications. Eur J Trauma Emerg Surg. 2019 Jun;45(3):445-453. doi: 10.1007/s00068-018-0916-9. Epub 2018 Feb 2. PMID 29396757
- [Background] Park S, Ahn J, Gee AO, Kuntz AF, Esterhai JL. Compartment syndrome in tibial fractures. J Orthop Trauma. 2009 Aug;23(7):514-8. doi: 10.1097/BOT.0b013e3181a2815a. PMID 19633461
- [Background] Zura R, Xiong Z, Einhorn T, Watson JT, Ostrum RF, Prayson MJ, Della Rocca GJ, Mehta S, McKinley T, Wang Z, Steen RG. Epidemiology of Fracture Nonunion in 18 Human Bones. JAMA Surg. 2016 Nov 16;151(11):e162775. doi: 10.1001/jamasurg.2016.2775. Epub 2016 Nov 16. PMID 27603155
- [Background] Sprague S, Bhandari M. An economic evaluation of early versus delayed operative treatment in patients with closed tibial shaft fractures. Arch Orthop Trauma Surg. 2002 Jul;122(6):315-23. doi: 10.1007/s00402-001-0358-3. Epub 2001 Dec 12. PMID 12136294
- [Background] Anandasivam NS, Russo GS, Swallow MS, Basques BA, Samuel AM, Ondeck NT, Chung SH, Fischer JM, Bohl DD, Grauer JN. Tibial shaft fracture: A large-scale study defining the injured population and associated injuries. J Clin Orthop Trauma. 2017 Jul-Sep;8(3):225-231. doi: 10.1016/j.jcot.2017.07.012. Epub 2017 Jul 24. PMID 28951639
- [Background] Rosa N, Marta M, Vaz M, Tavares SMO, Simoes R, Magalhaes FD, Marques AT. Intramedullary nailing biomechanics: Evolution and challenges. Proc Inst Mech Eng H. 2019 Mar;233(3):295-308. doi: 10.1177/0954411919827044. PMID 30887900
- [Background] Eveleigh RJ. A review of biomechanical studies of intramedullary nails. Med Eng Phys. 1995 Jul;17(5):323-31. doi: 10.1016/1350-4533(95)97311-c. PMID 7670691
- [Background] Donegan DJ, Akinleye S, Taylor RM, Baldwin K, Mehta S. Intramedullary Nailing of Tibial Shaft Fractures: Size Matters. J Orthop Trauma. 2016 Jul;30(7):377-80. doi: 10.1097/BOT.0000000000000555. PMID 26825491